CLINICAL TRIAL: NCT05010928
Title: Using Tea-based Mouthwash Relieve Stomatitis and Oral Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 202001919A3
Record Dates: First submitted 2021-08-09; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Stomatitis
Keywords: Stomatitis; oral ulcers; oral mucosa; tea; mouthwash
MeSH Terms: conditions — Stomatitis; Oral Ulcer | interventions — Mouthwashes; Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tea mouthwash group (Experimental)
  Interventions: Combination Product: mouthwash with tea
- Control group (No Intervention)

INTERVENTIONS:
Combination Product: mouthwash with tea — Using tea as a base, supplemented with licorice to make mouthwash to relieve stomatitis.
  Arms: Tea mouthwash group

SUMMARY:
The aim of this study is to use a tea-based mouthwash to relieve pain and discomfort in patients with stomatitis and ulcers.

DETAILED DESCRIPTION:
The objective of this study is to use tea as a base, supplemented with licorice to reduce bitterness and astringency, to make mouthwash, and use tea's antioxidant and anti-inflammatory properties to relieve the pain and discomfort of stomatitis and ulcer patients. This study will observe the difference between saliva and oral mucosal cells before and after treatment, to find the mechanism of effective treatment of stomatitis.

ELIGIBILITY:
Inclusion Criteria:

age over 20 years old, male or female

Exclusion Criteria:

patients with oral cavity cancer, oropharyngeal cancer, and active bacterial infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-26 (Estimated); Primary Completion 2024-11-26 (Estimated); Study Completion 2024-11-26 (Estimated)

PRIMARY OUTCOMES:
Xerostomia questionnaire (XQ) | 4 weeks
  Questionnaires for symptoms relief of dry mouth
Xerostomia Inventory (XI) | 4 weeks
  A multi-item approach to measuring dry mouth

SECONDARY OUTCOMES:
Rate of oral mucosa cells with angiotensin-converting enzyme 2 (ACE2) staining (+) | 4 weeks
  Immunohistochemistry stain for ACE2 protein

CONTACTS AND LOCATIONS:
Locations (1):
- Chiayi chang Gung Memorial Hospital, Chiayi City, Taiwan